CLINICAL TRIAL: NCT06706921
Title: Usefulness of Tumor Heterogeneity Assessment in Patients With MCRPC Undergoing Radioligand Therapy With 177LU-PSMA-617 Using Serial 18F-DCFPYL, 18F-FDG and 18F-Fluciclovine PET/CT Predicting Clinical Outcome
Brief Title: 18F-Fluciclovine PET/CT Impact on Predicting Clinical Outcome of 177Lu-PSMA-617 Therapy in Patients With Prostate Cancer
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Gholam Reza Berenji, MD, Attending Physician, VA Greater Los Angeles Healthcare System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1819674
Record Dates: First submitted 2024-10-22; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-09

CONDITIONS: Prostatic Neoplasms; Prostatic Neoplasms, Castration-Resistant; Metastatic Prostate Cancer; Male Urogenital Diseases; Prostatic Diseases; Urogenital Diseases, Male; Genital Diseases, Male; Neoplasms; Neoplasms by Site; Urogenital Neoplasms; Genital Neoplasms, Male
Keywords: Prostate cancer; PET/CT; Radioligand Therapy; Metastatic Castration-Resistant Prostate Cancer; PSMA PET
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Neoplasms, Castration-Resistant; Male Urogenital Diseases; Prostatic Diseases; Genital Diseases, Male; Neoplasms; Neoplasms by Site; Urogenital Neoplasms; Genital Neoplasms, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- 18F-Fluciclovine PET/CT (Experimental): Subjects receive 18F-Fluciclovine PET/CT scans.
  Interventions: Drug: 18F-Fluciclovine PET/CT Scan

INTERVENTIONS:
Drug: 18F-Fluciclovine PET/CT Scan — In this prospective study, an 18F-Fluciclovine PET/CT will be additionally obtained at baseline (pre-LuPSMA RLT), and after the 2nd, 4th, 6th LuPSMA RLT cycles.18F-Fluciclovine PET/CT will be acquired within 7 days from the PSMA PET.

SUMMARY:
This a single-center, prospective, exploratory study. Patients with metastatic castration-resistant prostate cancer (mCRPC) scheduled to undergo Lutetium labelled prostate-specific membrane antigen radioligand therapy (LuPSMA RLT) at the West Los Angeles VA (WLA-VA) will be imaged with a baseline F-18 fluorodeoxyglucose positron emission tomography/computed tomography 18F-FDG PET/CT and a 18F-DCFPyL PET/CT (18F-DCFPyL (2-(3-{1-carboxy-5-[(6-18F-fluoro-pyridine-3-carbonyl)-amino]-pentyl}-ureido)-pentanedioic acid)positron emission tomography/computed tomography , as per standard of care in our institution. All patients further undergo eventual follow-up prostate-specific membrane antigen positron emission tomography (PSMA PET) after the 2nd, 4th, and 6th LuPSMA RLT cycle. In this prospective study, an18F-Fluciclovine positron emission tomography/computed tomography ( Axumin PET/CT )will be additionally obtained at baseline (pre-LuPSMA RLT), and after the 2nd, 4th, 6th LuPSMA RLT cycles. Axumin PET/CT will be acquired within 7 days from the PSMA PET.

This study is open to Veterans only.

DETAILED DESCRIPTION:
The imaging analysis will consist in obtaining quantitative measurements of lesion uptake on the pre- and post-LuPSMA RLT (lesion and whole-body SUVmax, SUVmean and tumor volume) at each time point on all PET/CT scans. PET metrics at the lesion- and whole-body level will be compared among different PET radiopharmaceuticals at the same time point, and changes over time will be assessed.

All patients will be followed-up at our institution and clinical outcome will be correlated to the imaging analysis assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mCRPC scheduled to undergo LuPSMA RLT.
* Willingness to undergo multiple serial PET/CT scans pre- and post-LuPSMA RLT.
* Ability of providing written informed consent.

Exclusion Criteria:

* Less than 18 years-old at the time of radiopharmaceutical administration.
* Medical condition, serious concurrent illness, or other extenuating circumstance that, in the opinion of the Investigator, may significantly interfere with study procedures or compliance.
* Contraindications to LuPSMA RLT.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
18F-Fluciclovine PET/CT Impact on Predicting Clinical Outcome of 177Lu-PSMA-617 Therapy in Patients With Prostate Cancer | From enrollment to end of treatment at 34 weeks.
  Whole-body and lesion-level SUVmean, SUVmax. SUVmax, or maximum standardized uptake value, is a measurement used in positron emission tomography (PET) scans to quantify how much glucose a tumor is metabolizing.

SECONDARY OUTCOMES:
Usefulness of Tumor Heterogeneity Assessment in Patients in Patients With MCRPC Undergoing Radioligand Therapy With 177LU-PSMA-617 Using Serial 18F-DCFPYL, 18F-FDG and 18F-Fluciclovine PET/CT Predicting Clinical Outcome. | From enrollment to end of treatment at 34 weeks
  Tumor volume on FDG, Axumin and DCFPyL PET/CT. Tumor volume is the amount of space a tumor occupies, measured in cubic centimeters (cc).

OTHER OUTCOMES:
Usefulness of Tumor Heterogeneity Assessment in Patients in Patients With MCRPC Undergoing Radioligand Therapy With 177LU-PSMA-617 Using Serial 18F-DCFPYL, 18F-FDG and 18F-Fluciclovine PET/CT Predicting Clinical Outcome. | From enrollment to end of treatment at 34 weeks
  Percentage change in Whole-body and lesion-level SUVmean, SUVmax and tumor volume on FDG, Axumin and DCFPyL PET/CT pre- and post LuPSMA therapy. A "percentage change" refers to the calculated percentage difference between a initial value ( pre LuPSMA ) and a later measurement ( post LuPSMA ), essentially showing how much the tumor has grown or shrunk compared to its baseline size.

CONTACTS AND LOCATIONS:
Locations (1):
- VA Greater Los Angeles Healthcare System, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Study results are unknown at this time. The plan will be reevaluated once the results come in.